CLINICAL TRIAL: NCT05207215
Title: Use of Video Consultation, Computer Gaming and Self-help Home Exercises as Steps to Avoid Falls in the Elderly
Brief Title: Study on the Steps to Avoid Falls in the Elderly
Acronym: SAFETRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: SAFE TRIP
Record Dates: First submitted 2021-08-26; First posted 2022-01-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fall; Fall Prevention; Pre- Frail

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment randomized trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Video Conferencing (Active Comparator): Video conferencing is a 2-way interactive session that is enabled using telecommunication networks and the internet. The investigators will be working with 3rd party provider to create the video conferencing platform. Subjects can login to do SAFE exercises while physiotherapists monitor remotely. Subjects will complete two sessions per week (1hour for each session) for 12 weeks.
  Interventions: Other: Home Base Exercises
- Group B: Gamification (Active Comparator): Gamification refers to exercise-driven gaming, where games are developed with specifications/parameters that incorporate exercise movements. Currently, the investigators have an ongoing pilot study on game-assisted rehabilitation at SGH Physiotherapy Outpatient clinic and the exercise games are developed by an external company. The investigators will engage an external company to develop exercise games based on the exercises used in SAFE programme. Each game will have different difficulty levels to provide progressive training for subjects
  Interventions: Other: Home Base Exercises
- Group C: Self Guided (Active Comparator): Subjects in the self-guided exercise programme will be instructed to do SAFE exercises at least twice a week for an hour each by themselves.
  Interventions: Other: Home Base Exercises
- Group D: Self Guided (Placebo Comparator): Subjects in the self-guided exercise programme will be instructed to do SAFE exercises at least twice a week for an hour each by themselves.
  Interventions: Other: Home Base Exercises

INTERVENTIONS:
Other: Home Base Exercises — The study developed 3 approaches that innovate beyond the existing delivery modes of the SAFE programme, by developing means for providing an intervention that is functionally equivalent to the SAFE programme but can be implemented in a patient's home. These home approaches include: (a) video conferencing; (b) gamification; and (3) self-guided home exercise programme. The investigators' task is to focus on developing these 3 modes and evaluating each in a pilot context for participants upon discharge from the hospital.

SUMMARY:
This study focuses on administering home-based exercises which include balance, strength, endurance, and mobility training to pre-frail subjects via one of the 3 intervention arms. These evidence-based home exercises are performed two times a week for 12 weeks (3 months). A follow-up assessment will be conducted at the end of 9 months after 6 months maintenance phase.

DETAILED DESCRIPTION:
Falls are the most common morbid and expensive health condition involving older adults. The range of exercises included in the SAFE programme is designed to be adaptable to a wide range of physical functions targeting pre-frail older adults. The exact exercises will vary on the patients' functional status. However, all exercise sessions must include balance exercises that challenge the patient's balance during static activities, during movement and also may include challenges as the patient has divided attention (walking and talking, walking while carrying objects). Balance is first emphasised followed by strengthening exercises of the lower extremities. The improvement in walking, physical activity and endurance, is dependent on the patients' improvement in balance and strength. The overall design of the intervention is to develop and maintain functional mobility by targeting deficiencies in balance, strength, mobility, and endurance.

Despite efforts to provide exercises to improve patients' balance and strength to prevent falls, many do not comply with the programme upon discharge. To address this challenge, the investigators propose to conduct a pilot study that will employ novel approaches, using an evidence-based, person-centred falls prevention intervention (SAFE programme), which is sustainable and cost-effective for the general public in Singapore. These three interventions in the study include video conferencing, newly created exercise games (Gamification) and a self-guided home exercise programme.

A key aspect of the SAFE exercise programme is its simple yet structured series of exercises, with gradual progression, to improve balance, mobility and lower limb strength. It is important that subjects continually challenge themselves during the exercise sessions to promote ongoing improvement in physical function. An exercise stratification grid has been developed to help guide the subjects on the types of exercises and level of intensity, that will be appropriate for them. Performance level (as defined in the stratification grid) should be re-assessed weekly so as to track the progress of the subject i.e. once a subject has achieved the level of the specified exercise in a category, the participants will progress to the next level for the same category. In addition, the subjects will be encouraged to participate in walking both, as much and as far as possible, to improve their functional capacity. Therefore, the SAFE exercises are very appropriate to be used in the home setting.

140 pre-frail subjects discharged from SKH, SGH and OCH will be recruited for the study. Only those who meet the requirements criteria using the Ward PT Checklist will be randomised into the 3 intervention groups. All groups are required to exercise at least twice a week and complete the intervention over a 3-month period. Baseline, 3- and 9-months follow-up data will be collected by independent assessors. Outcome measures in 9 categories will be measured and compared across the 3 groups. These measures will be correlated to the subject's compliance to the intervention and effectiveness will be compared between the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60 years
* Singapore citizen or Permanent Resident
* With or without fall history in the last one year
* Short Physical Performance Battery (SPPB) >= 6
* Ability to provide informed consent
* Has not more than 1 major comorbidity (Heart attack, heart failure, cerebrovascular disease & cancer)
* Abbreviated Mental Test (AMT) >= 6
* Not referred for further active rehabilitation with a physiotherapist after discharge from hospital or outpatient care.

Exclusion Criteria:

* Patients who are advised by their physicians not to participate in physical activity sessions will be excluded from the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
To monitor the change of SPBB over the study period | Baseline, 3rd month and 9th month
  The SPBB will be captured at 3 time points (1st during the baseline, 2nd during the 3rd month post assessment and 3rd during the 9 month post assessment). Direct measurement will be taken by the assessor.

SECONDARY OUTCOMES:
Patient Demographic Profile | Baseline, 3rd month and 9th month
  The following will be collected Age, gender, ethnicity, marital status via an interview
Profile of the Caregiver | Baseline, 3rd month and 9th month
  This profile will be collected via an Interview
Health Status: Presence of diseases | Baseline, 3rd month and 9th month
  This information will be collected via an interview
Health Status: Lawton IADL | Baseline, 3rd month and 9th month
  This information will be collected via an interview
History & Attitude Towards Falls | Baseline, 3rd month and 9th month
  This information will be collected via an interview
Social Network & Social Isolation | Baseline, 3rd month and 9th month
  Variables for Lubben Social Network Scale (LSNS-6) are collected via interview.
Healthcare Utilisation | Baseline, 3rd month and 9th month
  The following variables are collected via interview:
  1. Number of visits by the participants to the Accident & Emergency Department
  2. Number of hospital admissions by the participants
  3. Number of visits by the participants to the General practitioner
Quality of Life Characteristics | Baseline, 3rd month and 9th month
  Variables for EQ-5D-5L are collected via interview.
Compliance of the different Intervention | Baseline, 3rd month and 9th month
  Variables for compliance are being collected via log book and weekly calls.

CONTACTS AND LOCATIONS:
Overall Officials: Celia IC Tan, PhD, Principal Investigator — SingHealth Services
Locations (1):
- Singapore General Hospital, Singapore, State *, Singapore

IPD SHARING:
Plan to Share IPD: No